CLINICAL TRIAL: NCT02378727
Title: CompuFlo® Assessment Study (COMPASS): A Randomized, Controlled, Parallel Group, Multicenter, Pivotal Study to Assess the Safety and Effectiveness of the Epidural Space Verification With the CompuFlo® Epidural Computer Controlled System
Brief Title: CompuFlo® Assessment Study for the Epidural Space Verification
Acronym: COMPASS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Milestone Scientific, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Diagnostic
Other Study IDs: EPI-INT14-01
Record Dates: First submitted 2015-02-23; First posted 2015-03-04 (Estimated); Last update posted 2016-07-06 (Estimated); Status verified 2016-06

CONDITIONS: Verification of Needle Tip Placement in the Lumbar Epidural Space

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A Standard Care Group (SCG) (Active Comparator): Standard Care Conventional Group (SCG): 158 subjects to receive lumbar epidural procedure with the loss of resistance syringe used to identify the epidural space
  Interventions: Device: Active: Comparator Loss Of Resistance Syringe
- Experimental Procedure Group (EPG). (Experimental): 158 of subjects to receive lumbar epidural procedure with the CompuFlo® Epidural System used to identify the epidural space
  Interventions: Device: Experimental: CompuFlo® Epidural System

INTERVENTIONS:
Device: Active: Comparator Loss Of Resistance Syringe — Lumbar epidural procedure utilizing Loss of Resistance Syringe
  Arms: A Standard Care Group (SCG)
Device: Experimental: CompuFlo® Epidural System — CompuFlo® Epidural is intended for use with an epidural needle for the verification of needle tip placement in the lumbar epidural space
  Arms: Experimental Procedure Group (EPG).

SUMMARY:
The purpose of this pivotal study is to demonstrate safety and effectiveness of the CompuFlo® Epidural Computer Controlled System (referred to hereafter as CompuFlo® Epidural) for the epidural space verification.

The CompuFlo® Epidural System is limited by federal law for investigational use only in United States of America and has received CE mark in European Union.

ELIGIBILITY:
Inclusion Criteria:

1. The Subject is at least 18 years of age at screening, but has not had their 91st birthday.
2. The Subject is required to have epidural procedure implemented as part of their standard medical treatment according to Principal Investigator assessment.
3. The Subject is willing to undergo the Informed Consent process prior to enrollment into this study.
4. The Subject is willing to participate in this study for at least 30 days after the epidural procedure implementation.
5. The Subject is willing to participate in this study for at least 3 days after the procedure.

Exclusion Criteria:

1. Contraindications for epidural procedure / anesthesia (circumstances where the risks associated with epidural procedures are higher than usual. These circumstances include, but are not limited to anatomical abnormalities, such as spina bifida or scoliosis, infection at or near the site of insertion, allergy to the anesthetic or intended drug, uncorrected hypovolemia, increased intracranial pressure etc.).
2. Patients presenting for emergency c-section or other emergencies.
3. Exclusive use of other treatments such as intravenous analgesia with opioids.
4. Prior back surgery in lumbar area that would prevent epidural access.
5. Preexisting neurological deficit that would interfere with dermatome identification.
6. The Subject observed seizure within 7 days prior to study enrollment.
7. Presumed and/or confirmed septic embolus.
8. The Subject has a skin condition (i.e., hemangioma, scleroderma, psoriasis, rash, open wound or tattoo) in their lumbar region greater than 4 cm2.
9. The Subject previously participated in another investigational drug or device trial within the preceding 4 weeks.
10. Severe co-existing or terminal systemic disease that limits life expectancy or may interfere with study procedures.
11. The Subject is otherwise determined by the Investigator to be medically unsuitable for participation in this study.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2015-01; Primary Completion 2016-07 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Primary Effectiveness Objective (successful performance of lumbar epidural procedure) | 1 week
  Primary study endpoint is successful performance of lumbar epidural procedure indicated by loss to temperature sensation bilateral either 1) (i) in at least one dermatome for the non-labor procedures procedures or (ii) in at least two dermatomes for women in labor two dermatomes*, based on a maximum of 3 attempts at epidural space identificationor 2) by correct spread of dye in the epidural space as observed by fluoroscopy for those patients for whom fluoroscopy is performed as a standard medical procedure to identify the exact spine level (landmarking) along with confirmatory contrast dye, based on a maximum of 3 attempts at epidural space identification This is a binary categorical (yes/no) endpoint.

CONTACTS AND LOCATIONS:
Overall Officials: Ralf Gebhard, MD, Study Chair — Professor of Anesthesiology Professor of Orthopedics and Rehabilitation Director, Division of Regional Anesthesia and Acute Perioperative Pain Management University of Miami-Miller School of Medicine
Locations (5):
- United States (5):
  - University of California Irvine, Irvine, California
  - Vitamed Research, Rancho Mirage, California
  - San Diego Pain Institute, San Diego, California
  - Northwestern Memorial Hospital, Chicago, Illinois
  - University of Texas Houston, Houston, Texas

IPD SHARING:
Plan to Share IPD: Undecided